CLINICAL TRIAL: NCT00205699
Title: Metabolic Effects of Antipsychotics in Children
Acronym: MEAC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NIMH; R01MH072912 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Results first posted 2018-06-15 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Aggression; Attention Deficit-Hyperactivity; Oppositional Defiant Disorder; Pervasive Development Disorders; Bipolar Disorder
Keywords: Antipsychotic treatment; Insulin action/secretion; Abdominal fat mass, total body fat; Aggression; Resting metabolic rates
MeSH Terms: conditions — Aggression; Oppositional Defiant Disorder; Child Development Disorders, Pervasive; Bipolar Disorder | interventions — Risperidone; Olanzapine; Aripiprazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- aripiprazole (Active Comparator): Participants in this group will be randomized to flexibly-dosed treatment with aripiprazole.
  Interventions: Drug: aripiprazole
- olanzapine (Active Comparator): Participants in this group will be randomized to flexibly-dosed treatment with olanzapine.
  Interventions: Drug: olanzapine
- risperidone (Active Comparator): Participants in this group will be randomized to flexibly-dosed treatment with risperidone.
  Interventions: Drug: risperidone

INTERVENTIONS:
Drug: risperidone — randomized to begin 12 week trial of risperidone
  Other Names: Risperdal
  Arms: risperidone
Drug: olanzapine — randomized to begin 12 week trial of olanzapine
  Other Names: Zyprexa
  Arms: olanzapine
Drug: aripiprazole — randomized to 12 week trial of aripiprazole
  Other Names: Abilify
  Arms: aripiprazole

SUMMARY:
The project aims to describe and compare the outcome of 12 weeks of prospective, randomized treatment with olanzapine, risperidone or aripiprazole on insulin action in skeletal muscle, liver and adipose tissue, abdominal fat mass, total body and fat-free mass, efficacy for symptoms of aggression and non-metabolic adverse events. Children aged 6-18 will be studied, exploring effects of stimulant therapy and age-related differences in vulnerability to treatment-induced adverse metabolic changes. Aims are addressed by measuring glucose and lipid kinetics with stable isotope tracers, body composition with dual energy x-ray absorptiometry and magnetic resonance imaging (MRI), and standardized assessments of efficacy and adverse events. Relevant data are critically needed to target clinical therapy and basic research, identify medical risks, and guide regulatory decisions in this vulnerable population.

DETAILED DESCRIPTION:
This randomized clinical trial assesses both the safety and efficacy of atypical antipsychotic agents in antipsychotic-naive aggressive children with various childhood psychiatric disorders during 12 weeks of prospective, randomized treatment with olanzapine, risperidone or aripiprazole.

Aim 1: To evaluate effects of selected antipsychotic treatments on insulin action in muscle (glucose disposal), liver (glucose production) and adipose tissue (lipolysis).

Aim 2: To evaluate effects of selected antipsychotic treatments on abdominal fat mass, total body fat and total fat-free mass.

ELIGIBILITY:
Inclusion Criteria:

* Aged 6-18 years
* Generally healthy and a score of ≥ 18 on the Aberrant Behavior Checklist in the context of one or more Axis I Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) childhood psychiatric disorders, including conduct disorder, oppositional defiant disorder, disruptive behavior disorder, autism, pervasive developmental disorder, attention deficit disorder, schizophrenia and bipolar affective disorders
* Children's Global Assessment Scale (CGAS) score ≤ 60
* Not previously treated with an antipsychotic; individual subjects with remote, brief prior antipsychotic exposure may be considered for enrollment by the PI on a case by case basis
* Patient assent and informed consent obtained from the parent or guardian
* No clinically significant (based on PI determination) changes in permitted medications (e.g., stimulants and selective serotonin reuptake inhibitors [SSRIs]) for approximately 1 month prior to Baseline evaluations

Exclusion Criteria:

* Active suicidality or primary dx of major depressive disorder
* Any lifetime use of antipsychotics or non-serotonin selective reuptake inhibitor (non-SSRI) anti-depressants
* The presence of any serious medical disorder, based on PI determination, that may confound the assessment of relevant biologic measures or diagnoses, including:

  * significant organ system dysfunction;
  * endocrine disease, including type 1 or type 2 diabetes mellitus;
  * coagulopathy;
  * anemia;
  * or acute infection.
* Subjects regularly taking any glucose lowering agent, lipid lowering agent, exogenous testosterone, recombinant human growth hormone, or any other endocrine agent that might confound substrate metabolism, oral glucocorticoids (glucocorticoid inhalants and nasal sprays are permitted), antihistamines, sedating antihistamines (non-sedating antihistamines such as but not limited to Claritin (loratadine) and Zyrtec (cetirizine) are permitted), and certain mood stabilizing agents, as some medications may themselves worsen or otherwise alter weight gain, glucose and lipid regulation or otherwise make it difficult to assess the effects of the antipsychotic alone; (note that exposure to many psychotropic agents including stimulants and SSRI's is permitted in order to maintain the generalizability of the sample);
* Intelligence quotient (IQ) < 70 (based on school records and/or evaluation by clinician)
* current substance abuse
* Past history or currently has dyskinesia
* Stimulant dosage significantly higher (per PI judgment)than the equivalent of approximately 2mg/kg/day methylphenidate equivalent dose.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 144 (Actual)
Dates: Start 2006-04 (Actual); Primary Completion 2011-03 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John W. Newcomer, MD, Principal Investigator — Florida Atlantic University and Washington University School of Medicine; Ginger Nicol, MD, Study Director — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, Psychiatry Dept., St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nicol GE, Yingling MD, Flavin KS, Schweiger JA, Patterson BW, Schechtman KB, Newcomer JW. Metabolic Effects of Antipsychotics on Adiposity and Insulin Sensitivity in Youths: A Randomized Clinical Trial. JAMA Psychiatry. 2018 Aug 1;75(8):788-796. doi: 10.1001/jamapsychiatry.2018.1088. PMID 29898210

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Post-enrollment screening for inclusion and exclusion criteria, e.g. for exclusionary conditions like diabetes mellitus.
Groups:
- Risperidone: 12 weeks of randomized treatment with flexibly dosed risperidone
- Olanzapine: 12 weeks of randomized treatment with flexibly dosed olanzapine
- Aripiprazole: 12 weeks of randomized treatment with flexibly dosed aripiprazole
Period: Overall Study
Arm/Group | Risperidone | Olanzapine | Aripiprazole
Started | 49 | 46 | 49
Completed | 46 | 40 | 43
Not Completed | 3 | 6 | 6
Not completed — Lost to Follow-up | 1 | 3 | 5
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 1
Not completed — Lack of Efficacy | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Risperidone: 12 weeks randomized, flexibly-dosed treatment with risperidone
- Olanzapine: 12 weeks randomized, flexibly-dosed treatment with olanzapine
- Aripiprazole: 12 weeks randomized, flexibly-dosed treatment with aripiprazole
- Total: Total of all reporting groups
Arm/Group | Risperidone | Olanzapine | Aripiprazole | Total
Number analyzed (Participants) | 49 | 46 | 49 | 144
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.32 (2.95) | 11.10 (2.52) | 11.60 (2.92) | 11.35 (2.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 18 | 15 | 46
  Male | 36 | 28 | 34 | 98
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 1 | 4
  Not Hispanic or Latino | 47 | 45 | 48 | 140
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 24 | 22 | 19 | 65
  Non-White | 25 | 24 | 30 | 79
Primary Diagnosis [Number; unit: participants]
  Attention Deficit Hyperactivity Disorder | 28 | 23 | 29 | 80
  Disruptive Behavior Disorder | 8 | 11 | 13 | 32
  Mood Disorder | 7 | 5 | 4 | 16
  Autism Spectrum Disorder | 3 | 4 | 3 | 10
  Psychosis | 2 | 2 | 0 | 4
  Obsessive Compulsive Disorder | 0 | 1 | 0 | 1
  Tourette Disorder | 1 | 0 | 0 | 1
Clinical Global Improvement (CGI)-Severity of Illness [Number; unit: participants]
  Moderately ill | 18 | 19 | 23 | 60
  Markedly ill | 31 | 26 | 23 | 80
  Severely ill | 0 | 1 | 3 | 4
Aberrant Behavioral Checklist Subscales [Mean (Standard Deviation); unit: units on a scale] — This instrument is a five-factor scale comprising 58 items in 5 sub scales. Items are scored on a scale of 0 (not a problem) to 3 (severe problem). Each sub scale score is the sum of items in the scale. The overall score is the sum of all items. Sub scales are Irritability (15 items, 0-45, clinical significance >18); Lethargy (16 items, min 0, max 48, clinical significance >9); Stereotypic Behavior; (7 items, 0 - 21, clinical significance >3) Hyperactivity, Noncompliance (16 items, 0-48, clinical significance >24); and Inappropriate Speech (4 items, 0-12, clinical significance >3).
  units on a scale
    Total | 88.03 (23.96) | 81.89 (21.55) | 83.53 (25.70) | 84.54 (23.82)
    Irritability/Aggression | 28.49 (5.53) | 28.17 (5.73) | 28.14 (6.27) | 28.27 (5.81)
    Lethargy | 16.57 (10.01) | 12.67 (8.15) | 14.61 (8.83) | 14.66 (9.12)
    Stereotypy | 5.54 (4.95) | 5.15 (4.42) | 4.29 (4.61) | 4.99 (4.67)
    Hyperactivity | 32.83 (9.68) | 32.11 (10.45) | 32.80 (10.88) | 32.59 (10.28)
    Inappropriate Speech | 4.60 (3.02) | 3.78 (2.71) | 3.69 (2.76) | 4.03 (2.85)
Clinical Global Assessment of Functioning [Mean (Standard Deviation); unit: units on a scale] — This instrument is a global measure of severity based on psychiatric symptomatology and impairment of adaptation in family, social, school, and work areas. On this scale 0 is worst, 100 is best, and ≤ 60 is definite clinical impairment.
  units on a scale | 51.71 (4.44) | 50.67 (5.44) | 50.88 (6.00) | 51.10 (5.31)
Number of Suspensions [Mean (Standard Deviation); unit: number of discrete school suspensions] — Population: Measure Analysis Population Description: The n's reported here represent complete data only.
  number of discrete school suspensions
    number analyzed (Participants) | 43 | 38 | 46 | 127
    (all) | 2.60 (4.11) | 2.71 (3.98) | 2.85 (4.18) | 2.72 (4.07)
On stimulant [Number; unit: participants]
  Yes | 29 | 21 | 22 | 72
  No | 20 | 25 | 27 | 72
On Selective Serotonin Reuptake Inhibitors (SSRI) [Number; unit: participants]
  Yes | 8 | 5 | 4 | 17
  No | 41 | 41 | 45 | 127
DEXA-measured body composition (%) [Mean (Standard Deviation); unit: percentage of body composition]
  DEXA Total % Fat | 26.25 (10.64) | 24.48 (10.19) | 26.23 (10.83) | 25.68 (10.52)
  DEXA Total % Lean | 70.30 (10.35) | 71.96 (9.96) | 70.32 (10.53) | 70.84 (10.25)
DEXA-measured body composition (kg) [Mean (Standard Deviation); unit: kilograms]
  DEXA Total Fat kg | 12.50 (9.53) | 10.46 (6.68) | 13.24 (10.40) | 12.10 (9.07)
  DEXA Total Lean kg | 30.38 (11.01) | 29.30 (9.83) | 31.98 (14.69) | 30.58 (12.04)
Baseline Insulin Stimulated % Change in Isotopomer Measurement during Week 0 Clamp [Mean (Standard Deviation); unit: % change during baseline clamp] — Population: Measure Analysis Population Description: Measure Analysis Population Description: The n's reported here represent complete data only.
  % change during baseline clamp
    % Change in Glucose Rate of Disappearance: number analyzed (Participants) | 42 | 34 | 41 | 117
    % Change in Glucose Rate of Disappearance | 166.26 (78.79) | 168.75 (82.09) | 156.49 (81.14) | 163.56 (80.06)
    % Change in Glucose Rate of Appearance: number analyzed (Participants) | 42 | 34 | 41 | 117
    % Change in Glucose Rate of Appearance | 83.19 (10.94) | 82.53 (9.90) | 82.70 (12.15) | 82.83 (11.01)
    % Change in Glycerol Rate of Appearance: number analyzed (Participants) | 42 | 34 | 41 | 117
    % Change in Glycerol Rate of Appearance | 55.59 (13.42) | 55.94 (15.08) | 50.46 (15.04) | 53.89 (14.59)
    Whole Body Sensitivity: number analyzed (Participants) | 47 | 44 | 48 | 139
    Whole Body Sensitivity | 12.96 (5.33) | 12.53 (4.47) | 12.87 (6.36) | 12.80 (5.44)
MRI-measured abdominal fat [Mean (Standard Deviation); unit: cm squared] — Population: The n's reported here represent complete data only.
  cm squared
    MRI Subcutaneous Fat: number analyzed (Participants) | 34 | 29 | 33 | 96
    MRI Subcutaneous Fat | 121.38 (123.05) | 86.17 (65.10) | 111.16 (94.16) | 107.23 (98.53)
    MRI Visceral Fat: number analyzed (Participants) | 34 | 30 | 33 | 97
    MRI Visceral Fat | 25.79 (18.45) | 19.37 (19.74) | 26.70 (24.14) | 24.11 (20.96)
    MRI Total Fat: number analyzed (Participants) | 34 | 29 | 33 | 96
    MRI Total Fat | 147.17 (137.36) | 106.09 (82.28) | 137.85 (116.24) | 131.56 (115.76)
Body Weight [Mean (Standard Deviation); unit: kilograms] | 45.49 (19.08) | 42.23 (13.81) | 47.94 (23.57) | 45.28 (19.34)
Waist Circumference [Mean (Standard Deviation); unit: centimeters] | 68.72 (13.47) | 65.87 (11.03) | 69.54 (15.50) | 68.09 (13.50)
Body Mass Index Percentile [Mean (Standard Deviation); unit: percentile] | 62.13 (29.70) | 58.38 (31.33) | 63.05 (30.12) | 61.25 (30.22)
Body Mass index z-score [Mean (Standard Deviation); unit: z-score] | 0.49 (1.12) | 0.30 (1.11) | 0.55 (1.13) | 0.45 (1.12)
Baseline fasting laboratory values (mg/dL) [Mean (Standard Deviation); unit: mg/dL]
  Fasting Glucose | 89.14 (8.81) | 87.48 (6.55) | 88.98 (6.16) | 88.56 (7.27)
  Total Cholesterol | 144.74 (28.88) | 137.09 (25.31) | 135.45 (28.34) | 139.14 (27.71)
  Triglycerides | 60.40 (33.00) | 60.98 (31.89) | 52.16 (23.13) | 57.78 (29.69)
  LDL Cholesterol | 79.53 (25.41) | 72.00 (24.56) | 72.82 (26.00) | 74.84 (25.40)
  Total Bilirubin | 0.37 (0.25) | 0.40 (0.18) | 0.33 (0.18) | 0.37 (0.21)
Baseline Fasting Laboratory Values (IU/L) [Mean (Standard Deviation); unit: IU/L]
  Alanine aminotransferase (ALT) | 18.10 (7.74) | 13.83 (4.20) | 15.53 (4.49) | 15.86 (5.96)
  Aspartate aminostransferase (AST) | 25.65 (7.10) | 23.26 (6.12) | 23.94 (6.78) | 24.31 (6.72)
  Alkaline Phosphatase | 209.33 (88.42) | 222.54 (75.69) | 206.41 (85.35) | 212.56 (83.19)
Baseline fasting laboratory values (g/dL) [Mean (Standard Deviation); unit: g/dL]
  Albumin | 4.02 (0.25) | 4.06 (0.27) | 4.05 (0.25) | 4.05 (0.25)
  Total Protein | 6.95 (0.46) | 6.90 (0.39) | 6.95 (0.34) | 6.94 (0.40)
High Sensitivity c-Reactive Protein (HS-CRP) [Mean (Standard Deviation); unit: mg/L] — Population: The n's reported here represent complete data only.
  mg/L
    number analyzed (Participants) | 48 | 46 | 48 | 142
    (all) | 1.61 (3.04) | 1.37 (3.04) | 1.12 (1.53) | 1.37 (2.62)
Fasting Insulin [Mean (Standard Deviation); unit: uU/mL] — Population: The n's reported here represent complete data only.
  uU/mL
    number analyzed (Participants) | 45 | 43 | 45 | 133
    (all) | 7.64 (5.85) | 6.24 (3.74) | 9.00 (8.68) | 7.65 (6.50)
Hemoglobin A1c [Mean (Standard Deviation); unit: %] | 5.46 (0.26) | 5.54 (0.34) | 5.54 (0.28) | 5.52 (0.29)

OUTCOME MEASURES:

1. Primary Outcome: Change in DEXA % Body Fat
Description: This study hypothesized that antipsychotic treatment would increase percent total body fat, as measured by whole body dual energy x-ray absorptiometry (DEXA), with larger adverse effects for olanzapine.
Time Frame: 12 weeks
Population: Modified Intent to Treat (ITT) sample with week 0 and week 12 data.
Measure: Mean (Standard Deviation); unit: percent body fat
Arm/Group | Risperidone | Olanzapine | Aripiprazole
Number analyzed (Participants) | 46 | 40 | 42
percent body fat | 1.81 (3.11) | 4.12 (3.10) | 1.66 (2.65)
Statistical Analysis 1: Comparison: Risperidone vs Olanzapine vs Aripiprazole; Primary analysis for change in DEXA % fat used a likelihood-based mixed-effects model using time (0, 6 and 12 weeks) and medication group as independent variables, with Toeplitz covariance structure specified, based on Bayesian information criteria (BIC). The null hypotheses were that there was no difference in the outcome over time (main effect of time) and that there were no differences between groups in the change over time (time by treatment condition); Test type: Superiority; p < 0.0001, Mixed Models Analysis — The p value refers to the time by treatment condition interaction. The a priori threshold for statistical significance in this planned primary test was p<0.05

2. Primary Outcome: Change in Insulin-stimulated Glucose Rate of Disappearance (Glucose Rd)
Description: This study hypothesized that antipsychotic treatment would decrease insulin sensitivity at muscle, as measured by the insulin-stimulated rate of disappearance of glucose (glucose Rd), with larger adverse effects for olanzapine.
Time Frame: 12 weeks
Population: Children ages 6-18 with a Diagnostic and Statistical Manual Text Revision (DSM-IV-TR) diagnosis and clinically significant aggression or irritability
Measure: Mean (Standard Deviation); unit: percentage of % change
Arm/Group | Risperidone | Olanzapine | Aripiprazole
Number analyzed (Participants) | 39 | 33 | 40
percentage of % change | 2.30 (83.91) | -29.34 (85.56) | -30.26 (65.46)
Statistical Analysis 1: Comparison: Risperidone vs Olanzapine vs Aripiprazole; Test type: Superiority; p = 0.07, ANCOVA

3. Secondary Outcome: Change in Insulin-stimulated Glycerol Rate of Appearance (Glycerol Ra)
Description: This study hypothesized that antipsychotic treatment would decrease insulin sensitivity at adipose tissue, as measured by the insulin-stimulated rate of disappearance of glycerol (glycerol Ra), with larger adverse effects for olanzapine.
Time Frame: 12 weeks
Population: Modified Intent to Treat (ITT) sample with week 0 and week 12 data.
Measure: Mean (Standard Deviation); unit: percentage of % change
Arm/Group | Risperidone | Olanzapine | Aripiprazole
Number analyzed (Participants) | 38 | 31 | 39
percentage of % change | -3.65 (17.23) | -8.29 (22.39) | 1.70 (16.79)
Statistical Analysis 1: Comparison: Risperidone vs Olanzapine vs Aripiprazole; Test type: Superiority; p = 0.27, ANCOVA

4. Secondary Outcome: Change in Insulin-stimulated Glucose Rate of Appearance (Glucose Ra)
Description: This study hypothesized that antipsychotic treatment would decrease hepatic insulin sensitivity, as measured by the rate of appearance of glucose (glucose Ra), with larger adverse effects for olanzapine.
Time Frame: 12 weeks
Population: Modified Intent to Treat (ITT) sample with week 0 and week 12 data.
Measure: Mean (Standard Deviation); unit: percentage of % change
Arm/Group | Risperidone | Olanzapine | Aripiprazole
Number analyzed (Participants) | 39 | 33 | 40
percentage of % change | -2.50 (7.61) | -6.57 (13.16) | -3.27 (9.27)
Statistical Analysis 1: Comparison: Risperidone vs Olanzapine vs Aripiprazole; Test type: Superiority; p = 0.17, ANCOVA

5. Secondary Outcome: Change in MRI-measured Visceral Abdominal Fat
Description: This study hypothesized that antipsychotic treatment would increase visceral abdominal fat, as measured by abdominal magnetic resonance imaging (MRI), with larger adverse effects for olanzapine.
Time Frame: 12 weeks
Population: Modified Intent to Treat (ITT) sample with week 0 and week 12 data.
Measure: Mean (Standard Deviation); unit: Change in cm-squared
Arm/Group | Risperidone | Olanzapine | Aripiprazole
Number analyzed (Participants) | 30 | 26 | 30
Change in cm-squared | 6.85 (10.99) | 10.73 (14.50) | 12.04 (15.11)
Statistical Analysis 1: Comparison: Risperidone vs Olanzapine vs Aripiprazole; Test type: Superiority; p = 0.29, ANCOVA

6. Secondary Outcome: Change in MRI-measured Subcutaneous Abdominal Fat
Description: This study hypothesized that antipsychotic treatment would increase subcutaneous abdominal fat, as measured by abdominal magnetic resonance imaging (MRI), with larger adverse effects for olanzapine.
Time Frame: 12 weeks
Population: Modified Intent to Treat (ITT) sample with week 0 and week 12 data.
Measure: Mean (Standard Deviation); unit: Change in cm-squared
Arm/Group | Risperidone | Olanzapine | Aripiprazole
Number analyzed (Participants) | 30 | 26 | 30
Change in cm-squared | 18.21 (22.27) | 34.27 (27.22) | 15.84 (19.02)
Statistical Analysis 1: Comparison: Risperidone vs Olanzapine vs Aripiprazole; Repeated measures ANCOVA was used to test for the main effect of time on the outcome, and to test for a time by treatment condition interaction that would indicate differences between groups in change over time in the primary outcome. The null hypotheses were that there was no difference in the outcome over time (main effect of time) and that there were no differences between groups in the change over time (time by treatment condition); Test type: Superiority; p < 0.003, ANCOVA
Statistical Analysis 2: Comparison: Risperidone vs Olanzapine; Test type: Superiority; p = 0.003, Contrast — Bonferroni correction for multiple comparisons was applied (p<0.05/4 = 0.0125); Contrasts based on the ANCOVA-derived time by treatment condition interaction
Statistical Analysis 3: Comparison: Olanzapine vs Aripiprazole; Test type: Superiority; p = 0.002, ANCOVA — Bonferroni correction for multiple comparisons was applied (p<0.05/4 = 0.0125); Contrasts based on the ANCOVA-derived time by treatment condition interaction

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the entire course of the study, April 2006 to July 2011 or 6 years and 3 months
Groups:
- Aripiprazole: Participants in this group were randomized to treatment with aripiprazole.
- Olanzapine: Participants in this group were randomized to treatment with olanzapine.
- Risperidone: Participants in this group were randomized to treatment with risperidone.
Arm/Group | Aripiprazole | Olanzapine | Risperidone
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/46 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/46 | 1/49
Other Adverse Events (participants affected / at risk) | 38/49 | 38/46 | 39/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aripiprazole (N=49) | Olanzapine (N=46) | Risperidone (N=49)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — About 2 months after starting Risperidone, participant had a complex partial seizure, later determined by a neurologist to be unrelated to study medication. Participant was restarted on the Risperidone.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole (N=49) | Olanzapine (N=46) | Risperidone (N=49)
Accidental Injury (Psychiatric disorders) | 3 | 3 | 5
Agitation (Psychiatric disorders) | 15 | 21 | 16
Anxiety (Psychiatric disorders) | 9 | 10 | 13
Constipation (Psychiatric disorders) | 1 | 2 | 7
Depression (Psychiatric disorders) | 1 | 5 | 4
Difficulty Concentrating (Psychiatric disorders) | 10 | 12 | 16
Drowsiness/Somnolence (Psychiatric disorders) | 11 | 10 | 8
Headache (Psychiatric disorders) | 4 | 4 | 5
Increased Appetite (Psychiatric disorders) | 18 | 31 | 15
Involuntary Movements (Psychiatric disorders) | 0 | 1 | 4
Restlessness (Psychiatric disorders) | 12 | 12 | 14
Runny Nose (Psychiatric disorders) | 6 | 1 | 1
Sleepiness (Psychiatric disorders) | 5 | 9 | 4
Thirst (Psychiatric disorders) | 1 | 3 | 1
Tiredness/Fatigue (Psychiatric disorders) | 6 | 6 | 2
Trouble Sleeping (Psychiatric disorders) | 4 | 3 | 8
Weight Gain (Psychiatric disorders) | 11 | 23 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Informed Consent Form: Child and Adult Consent (2010-10-18): https://cdn.clinicaltrials.gov/large-docs/99/NCT00205699/ICF_000.pdf
  • Informed Consent Form: Genetics Consent (2010-09-30): https://cdn.clinicaltrials.gov/large-docs/99/NCT00205699/ICF_001.pdf
  • Study Protocol (2018-03-22): https://cdn.clinicaltrials.gov/large-docs/99/NCT00205699/Prot_002.pdf
  • Statistical Analysis Plan (2018-03-28): https://cdn.clinicaltrials.gov/large-docs/99/NCT00205699/SAP_003.pdf